CLINICAL TRIAL: NCT06957483
Title: Acceptability, Fidelity, Safety and Preliminary Efficacy of a Sedentary Behaviour Intervention in Individuals With Spinal Cord Injury: a Pilot Study
Brief Title: Pilot Study of a Sedentary Behaviour Intervention for Individuals With a Spinal Cord Injury
Acronym: REACH-SCI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brunel University (Other)
Collaborators: Royal National Orthopaedic Hospital NHS Trust (Other)
Responsible Party: Principal Investigator, Dr Daniel Bailey, Reader in Sedentary Behaviour and Health, Brunel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 50038-NHS-Mar/2025-54084-2
Record Dates: First submitted 2025-04-23; First posted 2025-05-04 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injury
Keywords: Cardiovascular disease; Intervention; Paraplegia; Physical activity; Sedentary behaviour; Spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Cardiovascular Diseases; Paraplegia; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All participants will receive the REACH-SCI intervention in this single-arm study. The single arm will involve a wearable activity tracker, educational resources, goal setting, motivational support from a trained researcher, peer support and activity tools. The intervention period will be for eight weeks and will start after completion of all baseline measurements and provision of all intervention materials.
  Interventions: Behavioral: REACH-SCI (Reducing sedEntary Activities to improve Cardiovascular Health in individuals with a Spinal Cord Injury)

INTERVENTIONS:
Behavioral: REACH-SCI (Reducing sedEntary Activities to improve Cardiovascular Health in individuals with a Spinal Cord Injury) — The REACH-SCI intervention was co-designed with key stakeholders and aims to reduce and break up sedentary behaviour in individuals with paraplegia. The intervention will last eight weeks and involve (1) a wearable activity tracker to give reminders to break up sedentary behaviour, (2) education around what sedentary behaviour is, how to reduce and break up sedentary behaviour, and the benefits of doing so, (3) a goal setting worksheet related to sedentary behaviour, (4) one-to-one motivational support sessions to help set goals, review progress and give motivation, (5) peer support using a smartphone app, and (6) activity tools to support breaking up sedentary behaviour throughout the day.
  Other Names: REACH-SCI

SUMMARY:
Individuals with spinal cord injury have a greater risk of heart disease and stroke than non-disabled individuals. This might be partly because wheelchair users engage in high amounts of sedentary behaviour. A review found a lack of programmes aimed at reducing sedentary behaviour in individuals with paraplegia. This means we do not know how good these programmes are for reducing heart disease risk markers.

A programme to support reductions in sedentary behaviour has been co-designed with individuals with paraplegia, healthcare professionals, and people who support individuals with paraplegia in the community.

This study aims to evaluate the new programme to determine its acceptability, fidelity, safety and preliminary efficacy.

The Reducing sedEntary Activities to improve Cardiovascular Health in individuals with Spinal Cord Injury (REACH -SCI) intervention will last eight weeks and involve (1) a wearable activity tracker to give reminders to break up sedentary behaviour, (2) education around what sedentary behaviour is, how to reduce and break up sedentary behaviour, and the benefits of doing so, (3) a goal setting worksheet related to sedentary behaviour, (4) one-to-one motivational support sessions to help set goals, review progress and give motivation, (5) peer support using a group chat with other participants in a smartphone messaging app , and (6) activity tools (exercise bands and a handcycle) to support breaking up sedentary behaviour throughout the day.

Measurements of fatigue, pain, physical activity, sedentary behaviour, heart disease risk markers, wellbeing, anxiety, depression and quality of life will be taken at baseline before the programme starts and then again after the programme ends. Acceptability of the intervention and data collection procedures will be explored using semi-structured interviews and questionnaires.

DETAILED DESCRIPTION:
Background:

Individuals with a spinal cord injury are at a greater risk of heart disease and stroke than the general population. Many individuals with spinal cord injury sit for long periods due to being wheelchair users. Therefore, the increased risk of heart disease in this population may be partly linked to high levels of sedentary behaviour. However, the effects of sedentary behaviour interventions for individuals with paraplegia are not well understood. Also, interventions designed for non-disabled people are unlikely to be appropriate for individuals with paraplegia due to unique barriers linked to reliance on a manual wheelchair for mobility and other symptoms and limitations due to their injury.

A sedentary behaviour intervention tailored to the needs of individuals with paraplegia was co-designed with end users, healthcare professionals and key stakeholders . The primary aim of the study is to assess the acceptability, fidelity and safety of this co-designed intervention to reduce and break up sedentary behaviour in individuals with paraplegia. The main objectives are to:

* Explore participant acceptability of the intervention
* Explore fidelity of the intervention in the context of intervention components being delivered as planned, participant adherence and dosage
* Assess the safety of the intervention.

The secondary objectives are to:

* Evaluate participant engagement with the intervention components
* Explore the acceptability of data collection procedures
* Assess the feasibility of recruiting and retaining participants in the study
* Evaluate preliminary efficacy in the context of pre-post changes in sedentary behaviour, physical activity, cardiovascular disease biomarkers, psychosocial health and quality of life

Study design:

This pilot study will use a mixed-methods single-arm, pre-post design. After baseline measurements, all participants will receive the intervention. Measurements will be repeated eight weeks (end of intervention) following the start of the intervention period. Semi-structured interviews will also be undertaken by a subset of participants at eight weeks. Ethical approval has been granted from Brunel University of London College of Health, Medicine and Life Sciences Research Ethics Committee. Further approval will be sought from a National Health Service (NHS) Research Ethics Committee. The study will be undertaken in accordance with the Declaration of Helsinki and conducted and reported using the Consolidated Standards of Reporting Trials guidelines for feasibility and pilot trials.

Participant recruitment:

Participants will be recruited using purposive sampling in an effort to ensure the sample is representative of individuals throughout the SCI care pathway. Recruitment will take place in the community via disability sport and spinal cord injury pages on social media (e.g. X and Facebook), SCI charities (e.g. Spinal Injuries Association and Back-Up Trust), snowballing and participants from previous studies who have provided consent for being contacted about future research. Recruitment will also be through the London Spinal Cord Injury Centre, Royal National Orthopaedic Hospital NHS Trust. Potentially eligible patients will receive study information from a member of the care team during routine appointments, in-patient care and/or mail-out. Posters and leaflets containing study information will also be displayed within clinics and wards.

Intervention protocol:

The Reducing sedEntary Activities to improve Cardiovascular Health in individuals with Spinal Cord Injury (REACH-SCI) intervention will involve a wearable activity tracker, an educational booklet, goal setting, motivational support from a trained researcher, peer support from other participants and activity tools. The intervention period will be for eight weeks and will start after completion of all baseline measurements and provision of all intervention materials.

Wearable activity tracker:

Participants will be provided with a Garmin Vivoactive 5 (Garmin, Olathe, Kansas, USA) to be worn during the intervention. Verbal and printed guidance on how to set up, wear and use the device will be included. The device will be set up in Wheelchair Mode, which tracks pushes instead of steps and uses wheelchair-appropriate language.

The Garmin Vivoactive 5 provides reminders to break up sedentary behaviour with a haptic alert and notification to prompt physical activity after one hour of inactivity. Feedback on pushes, heart rate, calories burned and minutes spent in moderate- and vigorous-intensity physical activity is also provided through the wearable activity tracker interface and/or accompanying Garmin Connect smartphone app. Virtual badges are awarded to the participant for achieving personal push goals, sharing activities with friends in the app, completing challenges and doing different types of exercise. Streaks for consecutive days achieving personal push goals are also recorded within the app.

Participants can use their own wearable activity tracker if it has wheelchair mode, inactivity prompts, physical activity tracking and rewards to ensure all planned behaviour change techniques can be delivered.

Educational resources:

Participants will be provided with an educational booklet in both electronic and hard copy format. The booklet will cover (1) the definition of sedentary behaviour with examples of sedentary activities, (2) potential health benefits of reducing and breaking up sedentary behaviour, (3) ideas and suggestions to support reducing and breaking up sedentary behaviour including examples of how to involve family and friends, (4) how to set and review sedentary behaviour and physical activity goals and (5) a list of different charities, organisations and websites (with weblinks and contact information) who provide free or discounted exercise equipment, information and/or opportunities relating to physical activity and exercise.

Goal setting:

Participants will set short- and long-term goals related to sedentary behaviour and physical activity using a goal-setting worksheet and guidance from a trained researcher, as described below. Goals will be individualised, reflecting the amount and frequency at which participants aim to reduce or break up sedentary behaviour and, if viewed as appropriate, increase physical activity. Participants will be prompted and guided to estimate their current sedentary behaviour levels during both the first and final week of the intervention within the goal-setting worksheet. This will aid with reviewing progress toward their goals. Participants will also be encouraged and guided to set physical activity goals (e.g. daily pushes, intensity minutes) that could help contribute to reductions in sedentary behaviour within their wearable activity tracker to aid with tracking progress and feedback.

Motivational support sessions:

A researcher with training in motivational interviewing will support each participant in making behavioural changes. This will include support with setting individualised goals relating to sedentary behaviour and physical activity, reviewing goals and progress, and creating action plans. The one-to-one support sessions will be planned to take place via online video call or by phone, depending on participant preference. Three sessions will take place at approximately weeks 1, 3, and 5.

Peer support:

A peer support group will be set up by the research team in WhatsApp for those participating in the study to join if they wish. Participants will be encouraged to provide peer support and advice relating to sedentary behaviour and physical activity, and share experiences around taking part in the intervention. A member of the research team will send an initial message outlining the purpose of the group, ground rules and examples of what information could be shared. Reminder posts will be added each week to encourage continuous use of the chat.

Activity tools:

Participants will be provided with a pack of activity tools to use at home, which includes exercise bands of varying resistance and a portable hand cycle. Printed guidance around how and when to use the bands and hand cycle, including short, frequent bouts spread across the day to encourage breaks in sedentary behaviour, will be provided with the activity tools. The guidance will also include safety precautions around maintaining good shoulder health such as proper form and scheduling breaks.

Measurements:

At baseline, participant age, sex, ethnicity, comorbidities and spinal cord injury characteristics (neurological level, completeness, time since injury) will be collected to understand participant demographics. Study outcome measures include intervention acceptability, intervention fidelity, intervention safety, participant engagement, acceptability of data collection procedures, study feasibility, sedentary behaviour, physical activity, cardiovascular disease biomarkers and psychosocial health.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with self-reported paraplegia i.e. complete or incomplete SCI at T1 or below. Traumatic, non-traumatic, complete and incomplete SCI will all be eligible.
* At least 18 years of age.
* Self-report using a manual wheelchair as their primary mode of mobility inside and outside of the home.
* Able to travel to Brunel University of London to undertake study measurements.
* Access to use of a smartphone or tablet with internet access.
* Able to communicate in English at a level sufficient to understand the study, complete study measurements and engage fully with the intervention.
* Able to provide informed consent.
* Willing and able to provide fingertip blood samples and fast prior to measurement sessions.
* Able to independently transfer to a treatment couch and lay supine to undertake anthropometric measurements.

Exclusion Criteria:

* Self-reported heart condition, chest pain, dizziness, bone or joint problem, or any other condition that may be exacerbated by doing physical activity, as indicated via responses to the PAR-Q+.
* Self-reported history of uncontrolled autonomic dysreflexia in the past 12 months.
* Self-reported pregnancy.
* Currently participating in another research project that involves an intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Intervention acceptability | At intervention end (8 weeks)
  Following completion of the intervention, acceptability will be assessed via an adapted questionnaire with 5-point Likert scales and individual semi-structured interviews to explore constructs from the Theoretical Framework of Acceptability (TFA). The TFA assesses acceptability in the context of seven components (affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy), as well as overall intervention acceptability.
Intervention fidelity | From baseline to intervention end (8 weeks)
  Intervention fidelity will be assessed using a checklist to record each component being delivered as planned. This will include participants being provided with the wearable activity tracker, educational booklet, goal setting worksheet, exercise bands and portable hand cycle. Fidelity to the educational resource will be evaluated verbally in one-to-one motivational support sessions. Attendance at each motivational support session and duration of these sessions will be recorded. This will be in addition to a checklist for all planned aspects of the sessions being covered by the researcher delivering the intervention sessions.
Intervention safety - Adverse events | From baseline to intervention end (8 weeks)
  Safety of the intervention will be evaluated through adverse events (AE) experienced during the study. These will be self-reported at each data collection point, during contact with a facilitator as part of the intervention, and ad-hoc throughout the study by contacting a member of the research team via phone or email.
Intervention safety - Pain | Baseline and at intervention end (8 weeks)
  Safety will also be evaluated by measuring pain using the McGill Pain Questionnaire (MPQ), which is validated in individuals with SCI. Pain will be rated across 20 domains of pain using rating scales. Overall pain will be scored from 0 to 78, with a higher score representing worse levels of pain.
Intervention safety - Fatigue | Baseline and at intervention end (8 weeks)
  Safety will also be evaluated by measuring fatigue using the Modified Fatigue Impact Scale (MFIS), which is validated in individuals with SCI. Fatigue will be rated on a 5-point scale according to 21 domains of fatigue. Overall fatigue will be scored between 0 and 84, with a higher score representing worse levels of fatigue.

SECONDARY OUTCOMES:
Participant engagement | At intervention end (8 weeks)
  Intervention engagement will be assessed using a single questionnaire for participants to self-report how frequently they used the wearable activity tracker, educational resource booklet, goal-setting worksheets, peer support group chat and activity tools. Dose will also be measured through the same questionnaire where participants will report the time spent using each intervention component.
Acceptability of data collection procedures | At intervention end (8 weeks)
  Participant acceptability of the data collection procedures will be assessed via in-person semi-structured interviews.
Study feasibility | From recruitment to measurements taken at intervention end (8 weeks)
  Feasibility will be determined in the context of participant recruitment and retention rates and the proportion of missing data sets for daily sedentary time (proposed primary outcome for a definitive trial) and secondary outcomes.
Sedentary time | Baseline and in the final week of the intervention period
  A wrist-worn ActiGraph GT9X Link accelerometer will be used to collect activity data.
Physical activity | Baseline and in the final week of the intervention period
  A wrist-worn ActiGraph GT9X Link accelerometer will be used to collect activity data.
Body mass | Baseline and at intervention end (8 weeks)
  Total body mass will be measured using Marsden M-610 wheelchair scales.
Body mass index | Baseline and at intervention end (8 weeks)
  Body mass and height will be used to calculate body mass index, using the equation: kg/m^2.
Body fat mass | Baseline and at intervention end (8 weeks)
  Body fat mass will be measured using bioelectrical impedance analysis (Bodystat 1500).
Body fat percentage | Baseline and at intervention end (8 weeks)
  Body fat mass will be measured using bioelectrical impedance analysis (Bodystat 1500).
Waist circumference | Baseline and at intervention end (8 weeks)
  Waist circumference will be measured using an anatomical tape measure.
Diastolic blood pressure | Baseline and at intervention end (8 weeks)
  Blood pressure of the brachial artery will be measured using an A&D UA-611 automatic blood pressure monitor.
Systolic blood pressure | Baseline and at intervention end (8 weeks)
  Blood pressure of the brachial artery will be measured using an A&D UA-611 automatic blood pressure monitor.
Mean arterial pressure | Baseline and at intervention end (8 weeks)
  Mean arterial pressure will be measured via the following equation:
  (Diastolic X 2) + Systolic / 3
Fasting glucose | Baseline and at intervention end (8 weeks)
  Fasting fingertip capillary blood samples will be analysed using a CardioChek Plus automated analyser.
Fasting total cholesterol | Baseline and at intervention end (8 weeks)
  Fasting fingertip capillary blood samples will be analysed using a CardioChek Plus automated analyser.
Fasting HDL cholesterol | Baseline and at intervention end (8 weeks)
  Fasting fingertip capillary blood samples will be analysed using a CardioChek Plus automated analyser.
Total cholesterol to HDL cholesterol ratio | Baseline and at intervention end (8 weeks)
  Ratio will be calculated by dividing total cholesterol by HDL cholesterol.
Non-HDL cholesterol | Baseline and at intervention end (8 weeks)
  Outcome will be calculated by subtracting HDL cholesterol from total cholesterol.
Subjective wellbeing | Baseline and at intervention end (8 weeks)
  Office for National Statistics (2011) 4-item scale will be used to score subjective wellbeing between 0 and 10 in each domain. For the first three items, a higher score represents greater wellbeing. For the final item, a higher score represents worse wellbeing.
Anxiety | Baseline and at intervention end (8 weeks)
  Generalized Anxiety Disorder 7-item (GAD-7) questionnaire will be used to score anxiety between 0 and 3 in each domain. Overall anxiety will be scored between 0 and 21, with a higher score representing worse anxiety.
Depression | Baseline and at intervention end (8 weeks)
  Patient Health Questionnaire (PHQ-9) will be used to score depression between 0 and 3 across 9 domains. Overall depression will be scored between 0 and 27, with a higher score representing worse depression.
Health-related quality of life | Baseline and at intervention end (8 weeks)
  Modified 36-item Short-Form Health Survey (SF-36 walk wheel) will be used to score health-related quality of life across a scale in each of the 10 domains. Overall health-related quality of life will be scored between 0 and 100, with higher scores representing a better health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Bailey, PhD, Principal Investigator — Brunel University
Locations (1):
- Brunel University of London, Uxbridge, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Raw, anonymised data will also be made publicly available in an open research repository to ensure transparency and reproducibility, but only including data from participants who consent to this. All data will be saved on a password-protected laptop and University server.
Supporting Information: Study Protocol
Time Frame: Shared data will be available at study end following data analysis, after which there will be no time limit to gain access.
Access Criteria: Shared, anonymised data will be publicly available in an online open research repository.